CLINICAL TRIAL: NCT07397494
Title: Near Infrared Spectroscopy Imaging of Change in Tissue Oxygenation During a Provocative Leg Elevation Maneuver to Assess Peripheral Artery Disease: A Multicenter Study.
Brief Title: Near Infrared Spectroscopy Imaging of Change in Tissue Oxygenation to Assess Peripheral Artery Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Kent Imaging Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: K2024-02
Record Dates: First submitted 2026-01-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Peripheral Arterial Disease
Keywords: SnapshotNIR, PAD, NIR
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Suspected of PAD: subjects suspected of PAD
  Interventions: Other: Observational study only.

INTERVENTIONS:
Other: Observational study only. — Observational study only. All data collection will be completely observational and will not affect the patient care and treatment plan by any means.

SUMMARY:
This is a proof-of-concept study with exploratory objective to assess whether superficial tissue oxygenation patterns measured by Snapshot NIRS, in conjunction with the Provocative Elevation Maneuver of the Lower Extremity (PEMLE) and/or the Plantar Palmar Index (PPI), are associated with the severity of peripheral arterial disease (PAD) as determined by standard of care assessments and can be used to assess tissue oxygenation after revascularization, where applicable.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 21 and 99 years inclusive at the time of screening referred to the investigative site for further evaluation of known/suspected PAD.
* Subject has at least 1 intact forefoot.
* Can achieve leg positions as specified in the protocol to complete the study.
* Willing and able to provide written consent and adhere to protocol requirements

Exclusion Criteria:

* The subject is unwilling or unable to comply with the protocol (including but not limited to ability to tolerate leg lift) or scheduled appointments.
* The subject has had higher than trans metatarsal amputation on both limbs.
* Subjects who are pregnant, nursing or plan to become pregnant.
* For any reason as deemed appropriate by the Principal Investigator to be unsuitable for the study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be identified and enrolled through the PI's routine clinic population. Subjects who are identified for study participation will be screened for all eligibility requirements. Those meeting eligibility criteria for the study will have the study explained to them by the Principal investigator and have the opportunity to ask questions. An Informed Consent Form (ICF) will be signed prior to subjects undergoing any study procedures. Subjects will be encouraged to ask the study staff questions about the study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
To characterize superficial tissue oxygenation patterns, as measured by Snapshot NIRS, in patients with suspected or confirmed peripheral arterial disease (PAD). | baseline
  To characterize superficial tissue oxygenation patterns, as measured by Snapshot NIRS, in patients with suspected or confirmed peripheral arterial disease (PAD). PEMLE and PPI will be performed during the NIR assessment to support exploratory correlation with oxygenation patterns.

IPD SHARING:
Plan to Share IPD: No